CLINICAL TRIAL: NCT01494038
Title: A Phase IV Randomized Double-Blind Placebo-Controlled Trial to Evaluate the Safety of Immediate (Antepartum-Initiated) Versus Deferred (Postpartum-Initiated) Isoniazid Preventive Therapy Among HIV-Infected Women in High Tuberculosis (TB) Incidence Settings
Brief Title: Evaluating the Safety of Immediate Versus Deferred Isoniazid Preventive Therapy Among HIV-Infected Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P1078; 10732 (Registry Identifier: DAIDS ES); IMPAACT P1078
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2018-10

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Immediate INH Treatment) (Experimental): Women in Arm A received immediate, or antepartum-initiated, INH treatment. Women received INH at study entry through Week 28, then switched to placebo for INH treatment through Week 40 postpartum.
  Interventions: Drug: Isoniazid (INH); Drug: Placebo for isoniazid (INH)
- Arm B (Deferred INH Treatment) (Experimental): Women in Arm B received deferred, or postpartum-initiated, INH treatment. Women received placebo for INH at study entry through Week 12 postpartum, then switched to INH through Week 40 postpartum.
  Interventions: Drug: Isoniazid (INH); Drug: Placebo for isoniazid (INH)

INTERVENTIONS:
Drug: Isoniazid (INH) — 300-mg tablet once daily by mouth, either from entry through Week 28 antepartum (Arm A) or from Week 12 postpartum through Week 40 postpartum (Arm B)
Drug: Placebo for isoniazid (INH) — Placebo tablet once daily by mouth, either from Week 28 visit through Week 40 postpartum (Arm A) or from entry until Week 12 postpartum visit (Arm B)

SUMMARY:
Tuberculosis (TB) is a leading cause of death among HIV-infected persons in low-income settings and can be a serious complication for HIV-infected pregnant women and their infants. Isoniazid (INH) preventive therapy (IPT) is effective in preventing TB infection in HIV-infected adults, but the safety of IPT in pregnant women is unknown. This study evaluated the safety of IPT among HIV-infected pregnant women.

DETAILED DESCRIPTION:
TB disease is the most common HIV-related opportunistic infection and is a leading cause of death among HIV-infected persons in low-income settings. When TB occurs during or soon after pregnancy, it can cause complications for the mother as well as infant TB or death. Infant TB is very difficult to diagnose, and up to half of infant TB cases are caused by maternal TB. It has been shown that treatment for active TB is safe and effective during pregnancy and that IPT is safe and effective in preventing TB infection in HIV-infected adults. However, the safety of IPT in HIV-infected pregnant women is not known, especially in regard to its combination with highly active retroviral therapy (HAART). This study evaluated the safety of immediate (antepartum, or before delivery) versus deferred (postpartum, or after delivery) IPT among HIV-infected pregnant women in high TB incidence settings.

HIV-infected pregnant women were randomly assigned (1:1) to one of two arms: Arm A (immediate/antepartum INH) and Arm B (deferred/postpartum INH group). Women in both arms received oral prenatal multivitamins and pyridoxine (vitamin B6) once daily from study entry through Week 40 postpartum.

Study visits for women occurred at screening, entry, every 4 weeks until labor and delivery, at labor and delivery, and every 4 weeks after delivery until 48 weeks postpartum. Visits consisted of giving a medical history and undergoing a physical exam and blood collection; all visits through the delivery visit also included an obstetrical exam. Presence of HIV infection was documented at screening and a tuberculin skin test (TST) was administered at the delivery visit and at the Week 44 postpartum visit. Study visits for infants occurred at birth and at several time points through Week 48. These visits included a medical history, physical exam, and blood collection. Intensive pharmacokinetic (PK) samples, that is, samples taken at many different time points within a 24-hour test period, were collected from a small subset of women, one test period at antepartum and one at postpartum. Sparse PK samples, that is, samples taken at fewer time points within the test period, were collected on all women, once each at antepartum and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection, defined as positive results from two samples collected at different time points. All samples tested must be whole blood, serum, or plasma. More information on this criterion can be found in the protocol.
* Documented HIV treatment, according to World Health Organization (WHO) guidelines, for prevention of mother-to-child transmission (PMTCT) and standard of care for HIV infection
* Pregnant females age 18 years or older
* Pregnant females between greater than or equal to 13 and less than 18 who are able and willing to provide signed informed consent under local law or pregnant females unable to consent under local law whose parents/legal guardians provide consent or "minimum age of consent according to locally applicable laws or regulations"
* Pregnancy gestational age confirmed by best available method at site to be greater than or equal to 14 weeks through less than or equal to 34 weeks (34 weeks, 6 days)
* Weight greater than or equal to 35 kg at screening
* The following laboratory values obtained within 30 days prior to study entry:

  * Absolute neutrophil count (ANC) greater than or equal to 750 cells/mm^3
  * Hemoglobin greater than or equal to 7.5 g/dL
  * Platelet count greater than or equal to 50,000/mm^3
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT), alkaline phosphatase (ALT)/serum glutamic pyruvic transaminase (SGPT), and total bilirubin less than or equal to 1.25 times the upper limit of normal (ULN). (Note: If participant is taking atazanavir, direct bilirubin may be used to determine eligibility.)
* Intent to remain in current geographical area of residence for the duration of the study

Exclusion Criteria:

* Any woman with a positive TB symptom screen per WHO guidelines, including any one or more of the following: any cough, fever, self-reported weight loss, or night sweats. Note: If a potential participant is found to be negative for TB upon further testing, the participant may be rescreened for the study.
* Any positive acid-fast bacillus (AFB) smear, Xpert, or any other rapid TB screening test or culture from any site within the past 12 weeks, or chest radiograph (x-ray) with findings suggestive of active TB, or clinician suspects active TB
* Known exposure to AFB smear-positive active TB case within past 12 weeks prior to study entry
* Reported INH exposure (more than 30 days) in the past year prior to study entry
* Receipt of any TB or atypical mycobacteria therapy for more than 30 days in the past year
* Evidence of acute hepatitis, such as jaundice, dark urine (not concentrated urine), and/or acholic stools sustained for more than 3 days within 90 days prior to entry. More information on this criterion can be found in the protocol.
* Grade 1 or higher peripheral neuropathy. More information on this criterion can be found in the protocol.
* History of acute systemic adverse reaction or allergy to INH
* Known current heavy alcohol use (more than 2 drinks per week) or alcohol exposure that, in the investigator's opinion, would compromise participation and the outcome of this study
* Presence of new AIDS-defining opportunistic infection that has been treated less than 30 days prior to study entry
* Receipt of an investigational agent or chemotherapy for active malignancy within 30 days prior to study entry
* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise participation and the outcome of this study

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 956 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amita Gupta, MD, MHS, Study Chair — Johns Hopkins University
Locations (13):
- Botswana (2):
  - Gaborone CRS, Gaborone
  - Molepolole CRS, Gaborone
- Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince, Haiti
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- South Africa (3):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape
  - Fam-Cru Crs, Cape Town, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai, Thailand
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Zimbabwe (3):
  - Seke North CRS, Chitungwiza
  - St Mary's CRS, Chitungwiza
  - Harare Family Care CRS, Harare

REFERENCES:
- [Background] Akolo C, Adetifa I, Shepperd S, Volmink J. Treatment of latent tuberculosis infection in HIV infected persons. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD000171. doi: 10.1002/14651858.CD000171.pub3. PMID 20091503
- [Background] Zar HJ, Cotton MF, Strauss S, Karpakis J, Hussey G, Schaaf HS, Rabie H, Lombard CJ. Effect of isoniazid prophylaxis on mortality and incidence of tuberculosis in children with HIV: randomised controlled trial. BMJ. 2007 Jan 20;334(7585):136. doi: 10.1136/bmj.39000.486400.55. Epub 2006 Nov 3. PMID 17085459
- [Background] Cantwell MF, Snider DE Jr, Cauthen GM, Onorato IM. Epidemiology of tuberculosis in the United States, 1985 through 1992. JAMA. 1994 Aug 17;272(7):535-9. PMID 8046808
- [Derived] Gupta A, Singh P, Aaron L, Montepiedra G, Chipato T, Stranix-Chibanda L, Chanaiwa V, Vhembo T, Mutambanengwe M, Masheto G, Raesi M, Bradford S, Golner A, Costello D, Kulkarni V, Shayo A, Kabugho E, Jean-Phillippe P, Chakhtoura N, Sterling TR, Theron G, Weinberg A; IMPAACT P1078 TB APPRISE Study Team. Timing of maternal isoniazid preventive therapy on tuberculosis infection among infants exposed to HIV in low-income and middle-income settings: a secondary analysis of the TB APPRISE trial. Lancet Child Adolesc Health. 2023 Oct;7(10):708-717. doi: 10.1016/S2352-4642(23)00174-8. Epub 2023 Aug 24. PMID 37634517
- [Derived] Montepiedra G, Kim S, Weinberg A, Theron G, Sterling TR, LaCourse SM, Bradford S, Chakhtoura N, Jean-Philippe P, Evans S, Gupta A. Using a Composite Maternal-Infant Outcome Measure in Tuberculosis-Prevention Studies Among Pregnant Women. Clin Infect Dis. 2021 Aug 2;73(3):e587-e593. doi: 10.1093/cid/ciaa1674. PMID 33146706
- [Derived] Gupta A, Montepiedra G, Aaron L, Theron G, McCarthy K, Bradford S, Chipato T, Vhembo T, Stranix-Chibanda L, Onyango-Makumbi C, Masheto GR, Violari A, Mmbaga BT, Aurpibul L, Bhosale R, Mave V, Rouzier V, Hesseling A, Shin K, Zimmer B, Costello D, Sterling TR, Chakhtoura N, Jean-Philippe P, Weinberg A; IMPAACT P1078 TB APPRISE Study Team. Isoniazid Preventive Therapy in HIV-Infected Pregnant and Postpartum Women. N Engl J Med. 2019 Oct 3;381(14):1333-1346. doi: 10.1056/NEJMoa1813060. PMID 31577875
- See also: Manual for Expedited Reporting of Adverse Events to Division of AIDS (DAIDS), Version 2.0, January 2010 — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009) — http://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf?sfvrsn=6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected pregnant women and their infants, gestational age greater than 14 but less than 34 weeks, who reside in a high TB prevalence area. Recruited at participating medical clinics in those areas, a total of 13 sites in Haiti, India, Thailand, and in 5 countries in central and southern Africa. Recruitment from August 2014 to April 2016.
Groups:
- Arm A (Immediate INH Treatment): Women in Arm A received immediate, or antepartum-initiated, INH treatment. Women received INH at study entry through Week 28, then switched to placebo for INH treatment through Week 40 postpartum.
  Isoniazid (INH): 300-mg tablet once daily by mouth, from entry through Week 28 antepartum
  Placebo for isoniazid (INH): Placebo tablet once daily by mouth, from Week 28 visit through Week 40 postpartum
- Arm B (Deferred INH Treatment): Women in Arm B received deferred, or postpartum-initiated, INH treatment. Women received placebo for INH at study entry through Week 12 postpartum, then switched to INH through Week 40 postpartum.
  Isoniazid (INH): 300-mg tablet once daily by mouth, from Week 12 postpartum through Week 40 postpartum
  Placebo for isoniazid (INH): Placebo tablet once daily by mouth, from entry until Week 12 postpartum visit
Period: Overall Study
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Started | 477 | 479
Completed | 389 | 396
Not Completed | 88 | 83
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 18 | 20
Not completed — Withdrawal by Subject | 44 | 34
Not completed — Not able to get to clinic | 21 | 15
Not completed — Not willing to adhere to reqs | 2 | 9
Not completed — Death | 2 | 4

BASELINE CHARACTERISTICS:
Population: All women in study.
Groups:
- Arm B (Deferred INH Treatment): Women in Arm B received deferred, or postpartum-initiated, INH treatment. Women received placebo for INH at study entry through Week 12 postpartum, then switched to INH through Week 40 postpartum.
  Isoniazid (INH): 300-mg tablet once daily by mouth, from Week 12 postpartum through Week 40 postpartum (Arm B)
  Placebo for isoniazid (INH): Placebo tablet once daily by mouth, from entry until Week 12 postpartum visit (Arm B)
- Total: Total of all reporting groups
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment) | Total
Number analyzed (Participants) | 477 | 479 | 956
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [25 to 33] | 29 [24 to 33] | 29 [24 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 477 | 479 | 956
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 35 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 445 | 444 | 889
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Haiti | 8 | 15 | 23
  Botswana | 60 | 60 | 120
  Tanzania | 41 | 39 | 80
  South Africa | 91 | 91 | 182
  Uganda | 83 | 83 | 166
  Zimbabwe | 162 | 157 | 319
  Thailand | 15 | 18 | 33
  India | 17 | 16 | 33
Gestational age at entry [Count of Participants; unit: Participants]
  14 - <24 weeks | 161 | 160 | 321
  24 - 34 weeks | 316 | 319 | 635
CD4 Count [Count of Participants; unit: Participants] — Population: N=4 participants did not have baseline CD4 result available.
  Participants
    number analyzed (Participants) | 475 | 477 | 952
    < 350 cells/mm^3 | 118 | 114 | 232
    350 - <500 cells/mm^3 | 129 | 128 | 257
    500 - <650 cells/mm^3 | 95 | 105 | 200
    >= 650 cells/mm^3 | 133 | 130 | 263
Efavirenz-containing anti-retroviral (ARV) regimen [Count of Participants; unit: Participants]
  No | 72 | 70 | 142
  Yes | 405 | 409 | 814
Tuberculosis (TB) test result by Interferon-Gamma Release Assay (IGRA) [Count of Participants; unit: Participants] — Population: All enrolled participants with IGRA results available
  Participants
    number analyzed (Participants) | 470 | 472 | 942
    Positive | 139 | 144 | 283
    Negative | 301 | 297 | 598
    Indeterminate | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Combined Endpoint: Grade 3 or Higher Adverse Events (AEs) Related to Treatment, or AE Causing Discontinuation of Treatment
Description: Incidence rate, calculated by Mantel-Haenszel (MH), weighted by gestational age strata 1) gestational age at entry less than 24 weeks or 2) gestational age at entry greater than or equal to 24 weeks. AE's include laboratory results, signs/symptoms, or diagnoses; graded as per Division of AIDS (DAIDS) or by protocol-defined hepatotoxicity measures. Related to treatment indicates possibly, probably, or definitely related to INH or Placebo for INH as judged by Independent Endpoint Review Committee. Discontinuation refers to permanent discontinuation of study treatment.
Time Frame: Measured from study entry through Week 48 after birth
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Groups:
- Arm B (Deferred INH Treatment): Women in Arm B received deferred, or postpartum-initiated, INH treatment. Women received placebo for INH at study entry through Week 12 postpartum, then switched to INH through Week 40 postpartum.
  Isoniazid (INH): 300-mg tablet once daily by mouth, from Week 12 postpartum through Week 40 postpartum.
  Placebo for isoniazid (INH): Placebo tablet once daily by mouth, from entry until Week 12 postpartum visit.
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 15.03 | 14.93
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Non-Inferiority — Calculate the difference between the immediate arm incidence rate and the deferred arm incidence rate; if the upper bound of the 95% confidence interval is lower than a 5% difference in incidence rates, non-inferiority will be considered to be proven; Incidence rate difference = 0.10, 95% CI 2-sided [-4.77 to 4.98]

2. Secondary Outcome: Number of Mothers With a Fetal Death
Description: Fetal deaths include both stillbirths and spontaneous abortions; in case of a multiple birth, mothers who had at least one fetal death
Time Frame: Measured from study entry through end of pregnancy
Population: Mothers who had at least one live birth, stillbirth, or spontaneous abortion. One participant with outcome of induced abortion not included
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 459 | 466
Participants | 17 | 9
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = 0.093, Fisher Exact; mid-P adjustment

3. Secondary Outcome: Number of Mothers With a Fetus Small for Gestational Age
Description: Small for gestational age was determined by physician at site
Time Frame: Measured at delivery
Population: Measurement of small-for-gestational-age was deemed to be unreliable. Analysis not performed.
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Mothers With an Infant Born Prematurely
Description: Premature birth is defined as gestational age of < 37 weeks at delivery.
Time Frame: Measured at delivery
Population: Mothers who had at least one live birth
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 442 | 458
Participants | 48 | 40
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = 0.288, Fisher Exact; mid-P adjustment

5. Secondary Outcome: Number of Mothers With a Low Birth-weight Infant
Description: Low birth weight is defined as weight < 2500 mg
Time Frame: Measured on day of birth
Population: Mothers who had at least one live birth available to be weighed at time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 430 | 446
Participants
  Yes | 62 | 46
  No | 368 | 400
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = 0.073, Fisher Exact; mid-P adjustment

6. Secondary Outcome: Number of Mothers With an Infant With a Congenital Anomaly
Description: Includes congenital anomalies meeting the Metropolitan Atlanta Congenital Defects Program criteria.
Time Frame: Measured from study entry through Week 48 after birth
Population: Mothers who had at least one live birth able to be assessed between birth and 48 weeks after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 440 | 458
Participants
  Yes | 10 | 6
  No | 430 | 452
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = 0.264, Fisher Exact; mid-P adjustment

7. Secondary Outcome: Number of Mothers With an Adverse Pregnancy Outcome: Spontaneous Abortion, Stillbirth, Premature Birth, Low Birth Weight, or Congenital Anomaly
Description: In case of a multiple birth, mothers who had at least one adverse pregnancy outcome. Spontaneous abortion is intra-uterine fetal death prior to 20 weeks of gestational age; stillbirth, the same, >= 20 weeks; preterm delivery, < 37 weeks of gestational age; low birth weight, < 2,500 grams, and congenital anomalies meeting the Metropolitan Atlanta Congenital Defects Program criteria.
Time Frame: Measured from study entry through Week 48 after birth
Population: Mothers who had at least one live birth, stillbirth, or spontaneous abortion; participant with induced abortion is omitted, and whose babies were available for examination after birth (if born alive)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 449 | 460
Participants
  Yes | 106 | 78
  No | 343 | 382
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = 0.012, Fisher Exact; Mid-P adjustment

8. Secondary Outcome: Number of Infants With Grade 3 or Higher Clinical or Laboratory AE
Description: Laboratory, sign/symptom, or diagnoses graded as 3 or higher by DAIDS criteria.
Time Frame: Measured from study entry through Week 48 after birth
Population: Infants born alive
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
Participants | 193 | 196

9. Secondary Outcome: Number of Infants With Grade 3 or Higher Clinical or Laboratory AE Related to Treatment
Description: As before, but AE is judged to be possibly, probably, or definitely related to INH or Placebo for INH, by clinic medical staff
Time Frame: Measured from study entry through Week 48 after birth
Population: Infants born alive
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
Participants | 5 | 6

10. Secondary Outcome: Number of Infants Which Are HIV-infected
Description: HIV infection determined during follow-up period. Infection at birth or during breastfeeding
Time Frame: Measured from study entry through study Week 44
Population: Infants born alive
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
Participants
  Yes | 3 | 7
  No | 436 | 451
  Unknown | 6 | 6
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = 0.279, Fisher Exact; mid-P adjustment

11. Secondary Outcome: Number of Infants Hospitalized
Description: Hospitalization due to reasons other than birth
Time Frame: Measured from study entry through Week 48 after birth
Population: Infants born alive
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
Participants | 73 | 75
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; p = .893, Fisher Exact; mid-P adjustment

12. Secondary Outcome: Incidence Rate of TB Infection Among Mothers
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata. Probable or confirmed TB infection, as judged by Secondary Endpoint Review Committee
Time Frame: Measured from study entry to Week 48 after birth
Population: All participants enrolled without active TB at entry
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 478
events per 100 person-years | 0.60 | 0.59
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 0.01, 95% CI 2-sided [-0.94 to 0.96]

13. Secondary Outcome: Incidence Rate of Tuberculosis (TB) Among Infants
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata. Probable or confirmed TB, or congenital TB as defined using the Cantwell criteria (see reference), judged by the Secondary Endpoint Review Committee. Includes an infant death due to unknown cause.
Time Frame: Measured from study entry through Week 48 after birth
Population: Live-born infants of enrolled women
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
events per 100 person-years | 0.54 | 0.52
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 0.02, 95% CI 2-sided [-1.02 to 1.07]

14. Secondary Outcome: Incidence Rate of Infant Death
Description: Incidence rate was calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through Week 48 after birth
Population: Live-born infants of enrolled women
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
events per 100 person-years | 2.99 | 4.42
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -1.43, 95% CI 2-sided [-4.17 to 1.32]

15. Secondary Outcome: Incidence Rate of Maternal Deaths
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through Week 48 postpartum
Population: All participants enrolled without active TB at entry
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 478
events per 100 person-years | 0.40 | 0.78
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -0.39, 95% CI 2-sided [-1.33 to 0.56]

16. Secondary Outcome: Incidence Rate of Combined Endpoints: Maternal TB or Maternal Death
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through Week 48 after birth
Population: All participants enrolled without active TB at entry.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 478
events per 100 person-years | 1.00 | 1.38
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -0.38, 95% CI 2-sided [-1.72 to 0.97]

17. Secondary Outcome: Incidence Rate of Combined Endpoints: Infant TB or Infant Death
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through Week 48 after birth
Population: Live-born infants of enrolled women
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 445 | 464
events per 100 person-years | 2.99 | 4.68
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -1.69, 95% CI 2-sided [-4.48 to 1.1]

18. Secondary Outcome: Incidence Rate of Combined Endpoints: Maternal TB, Maternal Death, Infant TB, or Infant Death
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through Week 48 after birth
Population: Number of mother-infant pairs with at least one infant live birth and in which mother did not have active TB at entry.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 442 | 458
events per 100 person-years | 3.42 | 4.72
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -1.30, 95% CI 2-sided [-3.86 to 1.25]

19. Secondary Outcome: Incidence Rate of Combined Endpoint, Antepartum: Grade 3 or Higher AE Related to Treatment, or Discontinuation of Treatment Due to AE
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata
Time Frame: Measured from study entry through end of pregnancy
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 15.93 | 13.79
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 2.14, 95% CI 2-sided [-7.86 to 12.13]

20. Secondary Outcome: Incidence Rate of Combined Endpoint, up to 12 Weeks Postpartum: Grade 3 or Higher AE Related to Treatment, or Discontinuation of Treatment Due to AE
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through 12 weeks after birth
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 16.98 | 10.09
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 6.89, 95% CI 2-sided [-0.08 to 13.86]

21. Secondary Outcome: Incidence Rate, Antepartum, of Grade 3 or Higher AE
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through end of pregnancy
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 56.36 | 50.88
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 5.49, 95% CI 2-sided [-13.7 to 24.68]

22. Secondary Outcome: Incidence Rate, up to 12 Weeks Postpartum, of Grade 3 or Higher AE
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through 12 weeks postpartum
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 56.48 | 40.59
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 15.88, 95% CI 2-sided [2.11 to 29.65]

23. Secondary Outcome: Incidence Rate, Antepartum, of Hepatotoxicity, Defined by Protocol-specific Definition of Hepatotoxicity, Related to Treatment
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata. Protocol-specific definition of hepatotoxicity: Any one of the following: 1) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 5 times the upper limit of normal (ULN), where ULN is specified by the clinic physician; 2) Total bilirubin > 3 X ULN; 3) ALT greater than 3 X ULN and total bilirubin greater than 2 X ULN; or 4) ALT > 3 X ULN and persistent symptomatic clinical hepatitis
Time Frame: Measured from study entry through delivery
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 1.77 | 2.59
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -0.82, 95% CI 2-sided [-4.63 to 3]

24. Secondary Outcome: Incidence Rate, to 12 Weeks Postpartum, of Hepatotoxicity, Protocol-specific Definition, Related to Treatment
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata
Time Frame: Measured from study entry through 12 weeks postpartum
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 7.91 | 4.52
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 3.38, 95% CI 2-sided [-1.31 to 8.07]

25. Secondary Outcome: Incidence Rate, Antepartum, of Hepatotoxicity, Protocol-specific Definition, Any Cause
Description: Incidence rate calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through delivery
Population: All women enrolled.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 1.77 | 2.59
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -0.82, 95% CI 2-sided [-4.63 to 3]

26. Secondary Outcome: Incidence Rate, to 12 Weeks Postpartum, of Hepatotoxicity, Protocol-specific Definition, Any Cause
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through 12 weeks postpartum
Population: All women enrolled
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 8.37 | 4.98
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 3.39, 95% CI 2-sided [-1.46 to 8.25]

27. Secondary Outcome: Incidence Rate, Antepartum, of Hepatotoxicity, Defined by DAIDS, Related to Treatment
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata. Hepatotoxicity definition as defined by DAIDS AE grading criteria 1.0.
Time Frame: Measured from study entry through delivery
Population: All women.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 1.77 | 2.59
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -0.82, 95% CI 2-sided [-4.63 to 3]

28. Secondary Outcome: Incidence Rate, up to 12 Weeks Postpartum, of Hepatotoxicity, Defined by DAIDS, Related to Treatment
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata
Time Frame: Measured from study start through 12 weeks postpartum
Population: All women
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 7.91 | 4.52
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 3.38, 95% CI 2-sided [-1.31 to 8.07]

29. Secondary Outcome: Incidence Rate, Antepartum, of Hepatotoxicity, Defined by DAIDS, Any Cause
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study entry through delivery
Population: All women
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 1.77 | 2.59
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = -0.82, 95% CI 2-sided [-4.63 to 3]

30. Secondary Outcome: Incidence Rate, up to 12 Weeks Postpartum, of Hepatotoxicity, Defined by DAIDS, Any Cause
Description: Incidence rates calculated by Mantel-Haenszel, weighted by gestational age strata.
Time Frame: Measured from study start through 12 weeks postpartum
Population: All women.
Measure: Number; unit: events per 100 person-years
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
events per 100 person-years | 8.37 | 4.98
Statistical Analysis 1: Comparison: Arm A (Immediate INH Treatment) vs Arm B (Deferred INH Treatment); Test type: Superiority; Incidence rate difference = 3.39, 95% CI 2-sided [-1.46 to 8.25]

31. Secondary Outcome: Number of Mothers With Tuberculosis Resistant to INH
Description: Resistance to INH from isolates of Mycobacterium tuberculosis, as a percentage of mothers who develop culture-confirmed TB
Time Frame: Measured from study entry through Week 48 postpartum
Population: Mothers with culture-confirmed TB
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

32. Secondary Outcome: Number of Infants With Tuberculosis Resistant to INH
Description: Resistance to INH from isolates of Mycobacterium tuberculosis, as a percentage of infants who develop culture-confirmed TB
Time Frame: Measured from study entry through Week 48 after birth
Population: No infants had culture-confirmed TB
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Pharmacokinetic (PK) Parameter: Adjusted Mean of Area Under the Curve of Plasma Concentration Versus Time (AUC24h), for INH
Description: Pharmacokinetic parameter was estimated from population PK modeling fitted to the intensive PK data. AUC0-24h was predicted using population pharmacokinetic model using the NONMEM software program. A 2-compartment model with first-order absorption with transit compartment and first-order elimination with well-stirred liver model to capture hepatic clearance and first-pass extraction with 1 parameter (hepatic intrinsic clearance) was used,
Time Frame: Measured at antepartum (third trimester and >= 2 weeks after starting study drug) and week 16 postpartum (+/-) 4 weeks) while on active INH; blood samples were drawn pre-dose and at 1, 2, 4, 6, 8, and 12 hours post-dosing.
Population: Participants with intensive pharmacokinetic results while on active INH, who were established on INH.
Measure: Mean (95% Confidence Interval); unit: hour*mg/L
Groups:
- Fast Metabolizers: Those women having a genotype of fast INH metabolism.
- Intermediate Metabolizers: Those women having a genotype of intermediate INH metabolism.
- Slow Metabolizers: Those women having a genotype of slow INH metabolism.
Arm/Group | Fast Metabolizers | Intermediate Metabolizers | Slow Metabolizers
Number analyzed (Participants) | 5 | 15 | 12
hour*mg/L
  Third trimester of pregnancy | 3.63 [2.88 to 4.88] | 6.55 [5.31 to 7.88] | 21.6 [18.5 to 26.0]
  Week 16 postpartum | 4.25 [3.29 to 5.54] | 7.67 [6.49 to 9.18] | 25.3 [22.2 to 26.0]

34. Secondary Outcome: Pharmacokinetic (PK) Parameter: Adjusted Mean of Area Under the Curve (AUC24h), for EFV
Description: as for outcome 33
Time Frame: as for outcome 33
Population: Participants with intensive pharmacokinetic results while on active EFV and who were stabled on EFV-based ART.
Measure: Mean (95% Confidence Interval); unit: hour*mg/L
Groups:
- Fast Metabolizers: Those women with a phenotype of fast EFV metabolism.
- Intermediate Metabolizers: Those women with a phenotype of intermediate EFV metabolism.
- Slow Metabolizers: Those women with a phenotype of slow EFV metabolism.
Arm/Group | Fast Metabolizers | Intermediate Metabolizers | Slow Metabolizers
Number analyzed (Participants) | 3 | 10 | 8
hour*mg/L
  Third trimester of pregnancy | 38.5 [33.4 to 47.6] | 62.5 [51.4 to 94.9] | 153.02 [140.21 to 167]
  Week 16 postpartum | 46.9 [42.1 to 59.7] | 76.2 [61.1 to 111] | 186 [166 to 210]

35. Secondary Outcome: Agreement Between Interferon-gamma Release Assay (IGRA) TB Test and Tuberculin Skin Test (TST) Results, Women at Delivery
Description: IGRA done by Quantiferon Gold Test (QGIT). For women, TST is considered positive if greater than or equal to 5 mm
Time Frame: Measured at delivery
Population: Women tested for tuberculosis infection at delivery
Measure: Count of Participants; unit: Participants
Groups:
- Positive IGRA TB Test: Women who had positive IGRA TB test at delivery
- Negative IGRA TB Test: Women who had negative IGRA TB test at delivery
Arm/Group | Positive IGRA TB Test | Negative IGRA TB Test
Number analyzed (Participants) | 208 | 517
Participants
  Positive tuberculin skin test | 87 | 27
  Negative tuberculin skin test | 121 | 490
Statistical Analysis 1: Comparison: Positive IGRA TB Test vs Negative IGRA TB Test; Test type: Other — Measuring agreement between the tests; p < 0.0001, Chi-squared; McNemars test
Statistical Analysis 2: Comparison: Positive IGRA TB Test vs Negative IGRA TB Test; Test type: Other — Agreement between tests; Kappa coefficient = 0.42, 95% CI 2-sided [0.35 to 0.50]

36. Secondary Outcome: Agreement Between IGRA and TST TB Test Results, Infant
Description: The TST result was positive if greater than or equal to 10 mm in HIV-negative infants, or greater than or equal to 5 mm in HIV-positive infants.
Time Frame: Measured at week 44 after birth
Population: Infants with tuberculin tests performed at week 44 postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Positive IGRA Test: Infants with positive IGRA test at week 44 postpartum
- Negative IGRA Tuberculin Test: Infants with a negative IGRA test at 44 weeks postpartum
Arm/Group | Positive IGRA Test | Negative IGRA Tuberculin Test
Number analyzed (Participants) | 42 | 642
Participants
  Positive tuberculin skin test | 8 | 45
  Negative tuberculin skin test | 34 | 597
Statistical Analysis 1: Comparison: Positive IGRA Test vs Negative IGRA Tuberculin Test; Test type: Other — Agreement between tests; p = 0.22, Chi-squared; McNemar's test
Statistical Analysis 2: Comparison: Positive IGRA Test vs Negative IGRA Tuberculin Test; Test type: Other — Agreement between tests; Kappa coefficient = 0.11, 95% CI 2-sided [0.001 to 0.21]

37. Secondary Outcome: Agreement Between IGRA and TST TB Tests, Women at 44 Weeks Postpartum
Description: IGRA done by Quantiferon Gold Test (QGIT). For women, TST is considered positive if greater than or equal to 5 mm
Time Frame: Measured at Week 44 postpartum
Population: Women who were tested for tuberculosis infection at 44 weeks postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Positive IGRA TB Test: Women who had positive IGRA TB test at 44 weeks postpartum
- Negative IGRA TB Test: Women who had negative IGRA TB test at 44 weeks postpartum
Arm/Group | Positive IGRA TB Test | Negative IGRA TB Test
Number analyzed (Participants) | 227 | 479
Participants
  Positive tuberculin skin test | 100 | 20
  Negative tuberculin skin test | 127 | 459
Statistical Analysis 1: Comparison: Positive IGRA TB Test vs Negative IGRA TB Test; Test type: Other — Agreement between tests; p < 0.0001, Chi-squared; McNemar's test
Statistical Analysis 2: Comparison: Positive IGRA TB Test vs Negative IGRA TB Test; Test type: Other — Agreement between tests; Kappa coefficient = 0.46, 95% CI 2-sided [0.39 to 0.53]

38. Secondary Outcome: Number of Women by Level of Adherence to Prescribed Regimen, as Assessed by Self-report
Description: Adherence is the percentage of expected doses taken during the 28 week active treatment period, categorized as poor (<60%), reasonable (>= 60%, <80%), good (>=80%, <90%), or excellent (>= 90%). Measured by participant's self-report of doses taken within the last 3 days.
Time Frame: Adherence reported every 4 weeks during active treatment; study entry through week 28 for Arm A, week 12 postpartum through week 40 postpartum for Arm B
Population: All women enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
Participants
  Excellent adherence | 400 | 363
  Good adherence | 47 | 35
  Reasonable adherence | 15 | 8
  Poor adherence | 4 | 7
  Unknown | 11 | 66

39. Secondary Outcome: Number of Women by Level of Adherence to Prescribed Regimen, as Assessed by Pill Count
Description: Adherence is the percentage of expected doses taken during the 28 week active treatment period. Pill count: participants returned their prescription pill containers, and the remaining (unused) pills were counted.
Time Frame: as for outcome 38
Population: All enrolled women
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Immediate INH Treatment) | Arm B (Deferred INH Treatment)
Number analyzed (Participants) | 477 | 479
Participants
  Excellent adherence | 408 | 376
  Good adherence | 42 | 28
  Reasonable adherence | 8 | 6
  Poor adherence | 5 | 3
  Unknown | 14 | 66

ADVERSE EVENTS:
Time Frame: From study entry to study completion at week 48 postpartum or premature study discontinuation
Description: At entry, all diagnoses, signs/symptoms, and laboratory events were collected. Post-entry, all new diagnoses, signs/symptoms, or laboratory events of >= 3 and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade, were collected. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used. All eligible participants who initiated study treatment and their live-born infants are included.
Groups:
- Mother/Immediate INH: Women in Arm A received immediate, or antepartum-initiated, INH treatments. Women received INH at study entry through Week 28, then switched to placebo for INH treatment through Week 40 postpartum.
  Isoniazid (INH): 300-mg tablet once daily by mouth, from entry through Week 28 antepartum
  Placebo for isoniazid (INH): Placebo tablet once daily by mouth, from Week 28 visit through Week 40 postpartum.
- Mother/Deferred INH: Women in Arm B received deferred, or postpartum-initiated, INH treatment. Women received placebo for INH at study entry through Week 12 postpartum, then switched to INH through Week 40 postpartum.
  Isoniazid (INH): 300-mg tablet once daily by month, from Week 12 postpartum through Week 40 postpartum.
  Placebo for isoniazid (INH): Placebo tablet once daily by mouth, from entry until Week 12 postpartum visit.
- Infant/Immediate INH: Infants born alive to mothers on arm A (Immediate INH).
- Infant/Deferred INH: Infants born alive to mothers on Arm B (Deferred INH).
Arm/Group | Mother/Immediate INH | Mother/Deferred INH | Infant/Immediate INH | Infant/Deferred INH
All-Cause Mortality (participants affected / at risk) | 2/477 | 4/479 | 11/445 | 17/464
Serious Adverse Events (participants affected / at risk) | 71/477 | 69/479 | 86/445 | 91/464
Other Adverse Events (participants affected / at risk) | 438/477 | 449/479 | 417/445 | 430/464
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mother/Immediate INH (N=477) | Mother/Deferred INH (N=479) | Infant/Immediate INH (N=445) | Infant/Deferred INH (N=464)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemorrhagic disease of newborn (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Choledochal cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Congenital cytomegalovirus infection (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Exomphalos (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 2 | 1
Fever neonatal (General disorders) | 0 | 0 | 1 | 0
Macrosomia (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 3
Sudden infant death syndrome (General disorders) | 0 | 0 | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 4 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 3 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Rhesus incompatibility (Immune system disorders) | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Ascariasis (Infections and infestations) | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 3 | 5
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 3 | 3 | 6
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Haemophilus sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Herpangina (Infections and infestations) | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Parvovirus B19 infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 8 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 2 | 4
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Postpartum sepsis (Infections and infestations) | 1 | 2 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 2 | 2
Sepsis neonatal (Infections and infestations) | 0 | 0 | 11 | 16
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 7 | 5 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Induced abortion failed (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Convulsion neonatal (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Hypocalcaemic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 12 | 9 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 5 | 5 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 3 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 3
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 8 | 2 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 10 | 12
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 | 6 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 5 | 0 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Uterine inversion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Uterine atony (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 3
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 3
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 5
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mother/Immediate INH (N=477) | Mother/Deferred INH (N=479) | Infant/Immediate INH (N=445) | Infant/Deferred INH (N=464)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 36 | 41
Abdominal pain (Gastrointestinal disorders) | 24 | 15 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 37 | 25 | 79 | 83
Pyrexia (General disorders) | 12 | 11 | 51 | 57
Conjunctivitis (Infections and infestations) | 17 | 14 | 29 | 26
Gastroenteritis (Infections and infestations) | 25 | 20 | 58 | 50
Oral candidiasis (Infections and infestations) | 1 | 1 | 25 | 24
Upper respiratory tract infection (Infections and infestations) | 15 | 23 | 45 | 48
Urinary tract infection (Infections and infestations) | 55 | 51 | 2 | 2
Vulvovaginal candidiasis (Infections and infestations) | 52 | 47 | 0 | 0
Alanine aminotransferase increased (Investigations) | 187 | 206 | 31 | 31
Aspartate aminotransferase increased (Investigations) | 141 | 151 | 9 | 2
Blood alkaline phosphatase increased (Investigations) | 12 | 26 | 2 | 1
Blood glucose decreased (Investigations) | 144 | 128 | 1 | 1
Blood glucose increased (Investigations) | 40 | 47 | 0 | 0
Haemoglobin decreased (Investigations) | 199 | 191 | 353 | 365
Neutrophil count decreased (Investigations) | 81 | 87 | 270 | 264
Platelet count decreased (Investigations) | 22 | 10 | 23 | 26
Weight decreased (Investigations) | 96 | 97 | 15 | 12
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 23 | 23
Growth failure (Musculoskeletal and connective tissue disorders) | 0 | 0 | 47 | 38
Neuropathy peripheral (Nervous system disorders) | 94 | 109 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 35 | 66 | 87
Hypertension (Vascular disorders) | 40 | 37 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT01494038/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT01494038/SAP_000.pdf